CLINICAL TRIAL: NCT02899390
Title: Adaptation and Evaluation of a Diabetes Prevention Program About Parameters of Obesity, Physical Activity and Biochemical Parameters in Adults of the Yaqui Tribe of Hermosillo, Sonora at Risk of Diabetes
Brief Title: Diabetes Prevention Program in Adults of the Yaqui Tribe of Hermosillo, Sonora at Risk of Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Investigación en Alimentación y Desarrollo A.C. (Other)
Collaborators: Universidad de Sonora (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CentroIAD
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Prediabetes; Obesity; Overweight
MeSH Terms: conditions — Prediabetic State; Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle Intervention (Experimental): All the participants will be offered group and individual sessions to help them accomplish weight loss and also increase physical activity.
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention — Before implementation of the National Diabetes Prevention Program, adaptations will be made in order to be culturally acceptable in the community taking in consideration the type of food they eat and their activities in the population.
  The lifestyle intervention will be implemented by group and individual sessions and is aimed at achieving a 7% loss weight from baseline and 150 minutes per week of physical activity. Sessions will be held weekly in a period of 6 months. Individual sessions consist in nutritional counseling according to energy needs and food preferences of each participant.

SUMMARY:
Diabetes is a major non communicable chronic diseases in the world. It occupies the fourth or fifth leading cause of death in most high-income countries and there is strong evidence that has epidemic proportions in many developing countries, including Mexico. Like diabetes, prediabetes is associated with obesity and insulin resistance, thus promoting a lifestyle with healthy eating and physical activity can reduce weight and in turn the risk of diabetes.

Several studies have shown that it is possible to prevent or delay the development of type 2 diabetes through a lifestyle intervention based on diet and physical activity. The National Diabetes Prevention Program is a study based on the Diabetes Prevention Program conducted in real-world conditions.

It is known that the acculturation of some ethnic groups has led to the increase in certain chronic degenerative diseases due to increased associated risk factors. The rural Yaqui tribe has a high prevalence of overweight, obesity, high triglycerides and type 2 diabetes. In addition to the rural Yaqui tribe there is another settlement of this tribe in the city of Hermosillo Sonora. Information on the health of this ethnic group is limited, however, it is known that being seated in an urban setting with an obesogenic lifestyle, which has been shown to have serious health effects in other populations, suggesting a high prevalence chronic non-communicable diseases such as obesity, type 2 diabetes and hypertension at this ethnic group.

The present study is a translational research clinical trial to evaluate the effectiveness of the National Diabetes Prevention Program to improve obesity parameters (weight, BMI, waist circumference) and increase physical activity in adults who are at risk of diabetes in the Yaqui tribe established in Hermosillo, Sonora.

DETAILED DESCRIPTION:
The present project wants to know if a diabetes prevention program can reduce the risk of developing diabetes in adults at risk of the Yaqui tribe established in Hermosillo, through the loss of weight and physical activity, all these with an intensive lifestyle intervention program that provide them the benefits of a healthy nutrition and physical activity.

The hypothesis is that a lifestyle intervention program addressed to adults in the Yaqui tribe, established in Hermosillo at risk of diabetes can significantly decrease the parameters of obesity in a period of 6 months and increase physical activity in the same time period.

ELIGIBILITY:
Inclusion Criteria:

* Being part of the Yaqui tribe established in Hermosillo, Sonora.
* Age 20 years and less than 65
* FINDRISC score of 12 or higher
* Desire of participate
* Sign up the consent form

Exclusion Criteria:

* Diabetes diagnosis or another chronic disease
* Have been suffered a myocardial infarction in the last 6 months
* Cardiovascular disease
* Be seriously ill
* Use of medication that alter glucose tolerance
* Use of medicaments to lost weight
* Present conditions that affect their participation in the study (use of drugs or inability to exercise

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Body weight change | After 16 weekly sessions

SECONDARY OUTCOMES:
Change in Body Mass Index | After 16 weekly sessions
Change in waist circumference | After 16 weekly sessions
Change in body fat percentage | After 16 weekly sessions
Change in systolic and diastolic blood pressure | After 16 weekly sessions
Change in fasting glucose | After 16 weekly sessions
Change in total cholesterol | After 16 weekly sessions
Change in LDL-cholesterol | After 16 weekly sessions
Change in triglycerides | After 16 weekly sessions
Change in fasting insulin | After 16 weekly sessions
Change in the Beck Depression Inventory score | After 16 weekly sessions
Change in the Short Form-36 Health Survey score | After 16 weekly sessions
Change in the Perceived Stress Scale (PSS) -14 score | After 16 weekly sessions

CONTACTS AND LOCATIONS:
Overall Officials: Julián Esparza-Romero, Ph.D., Principal Investigator — Centro de Investigación en Alimentación y Desarrollo
Locations (3):
- Mexico (3):
  - Centro de Investigación en Alimentación y Desarrollo, Hermosillo, Sonora
  - Centro de Salud Urbano Los Naranjos, Hermosillo, Sonora
  - Elementary School Lázaro Mercado, Hermosillo, Sonora

IPD SHARING:
Plan to Share IPD: Undecided